CLINICAL TRIAL: NCT04004286
Title: Defense and Veterans Center for Integrative Pain Management (DVCIPM)Pain Registry Biobank
Brief Title: Defense and Veterans Center for Integrative Pain Management (DVCIPM) Pain Registry Biobank
Acronym: PRBiobank
Status: Recruiting | Type: Observational
Sponsor: Defense and Veterans Center for Integrative Pain Management (Other)
Responsible Party: Sponsor
Other Study IDs: 900405
Record Dates: First submitted 2019-06-13; First posted 2019-07-02 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Pain
Keywords: Pain PASTOR Biobank
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood specimens and saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This Pain Registry Biobank is a prospective cohort design study whereby data (PASTOR survey, blood and saliva specimens, clinical data) is collected from participants in a longitudinal fashion with continual enrollment.

DETAILED DESCRIPTION:
The Defense and Veterans Center for Integrative Pain Management (DVCIPM) established a clinical data registry and tissue biobank (pain registry/biobank) for the advancement of pain-related research. This Pain Registry Biobank will address the complexity of pain by utilizing the Pain Assessment Screening Tool & Outcomes Registry (PASTOR), a thorough biopsychosocial assessment that extends beyond a single-item pain rating scale. PASTOR is an assessment battery that includes several Patient Reported Outcomes Measurement Information System (PROMIS) scales developed by the National Institutes of Health (NIH) and other important scales that span physical, psychological, social, and behavioral aspects of pain and pain-related treatments. As a uniform assessment system, PASTOR also mitigates a significant challenge in pain-related research, the lack of standardized, cross-study outcomes. Additionally, the richness of PASTOR data matched with biological samples allows future researchers to address significant research gaps and enhance health care for service members, veterans, and civilians.

ELIGIBILITY:
Inclusion Criteria:

* Eligibile for care within the Military Healthcare System
* Able and willing to provide written consent

Exclusion Criteria:

* Cannot understand English

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Male and female military health care beneficiaries age 18 years and older presenting for an appointment care at WRNMMC
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2050-02 (Estimated); Study Completion 2050-02 (Estimated)

PRIMARY OUTCOMES:
Pain Registry: PASTOR survey | Up to 30 years
  a thorough biopsychosocial assessment computer adaptive screening tool that extends beyond a single-item pain rating scale. PASTOR is an assessment battery that includes several Patient Reported Outcomes Measurement Information System (PROMIS) scales developed by the National Institutes of Health (NIH) and other important scales that span physical, psychological, social, and behavioral aspects of pain and pain-related treatments.
Pain Registry: Blood specimens | Up to 30 years
  43 ml of blood collected and processed for storage from EDTA, BDP 100, PAXgene RNA, and DNA blood collection tubes
Pain Registry: Saliva | Up to 30 years
  up to 10ml of saliva, collected in 2ml cryovials.

CONTACTS AND LOCATIONS:
Overall Officials: Harold J Gelfand, MD, Principal Investigator — Defense and Veterans Center for Integrative Pain Management
Locations (2):
- United States (2):
  - Naval Medical Center San Diego, San Diego, California
  - Walter Reed National Military Medical Center, Bethesda, Maryland

DOCUMENTS (1):
  • Informed Consent Form (2020-02-01): https://cdn.clinicaltrials.gov/large-docs/86/NCT04004286/ICF_000.pdf